CLINICAL TRIAL: NCT06028750
Title: Accuracy of Dental Implant Placement Using Dynamic Navigation or the Freehand Method: a Randomized Controlled Clinical Trial in Novice Operators
Brief Title: Dynamic Navigation vs. the Freehand Method
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Barcelona (Other)
Responsible Party: Principal Investigator, Octavi Camps-Font, Associate Professor of Oral Surgery, University of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: RCT X-GUIDE (50/2022)
Record Dates: First submitted 2023-05-08; First posted 2023-09-08 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Dental Implants
Keywords: Dynamic computer assisted implant surgery

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Freehand (Active Comparator): Nobel Replace Conical Connection® placed freehand
  Interventions: Procedure: Freehand
- X-Guide guided surgery system (X-Nav Technologies®, Pennsylvania, USA) (Experimental): Nobel Replace Conical Connection® placed using the X-Guide guided surgery system (X-Nav Technologies®, Pennsylvania, USA)
  Interventions: Procedure: Dynamic Computer Assisted Surgery

INTERVENTIONS:
Procedure: Dynamic Computer Assisted Surgery — Surgical navigation system (X-Guide guided surgery system) Navigation system X-Guide
  Other Names: Dynamic Navigation; Navigated surgery
  Arms: X-Guide guided surgery system (X-Nav Technologies®, Pennsylvania, USA)
Procedure: Freehand — Freehand implant placement
  Arms: Freehand

SUMMARY:
The purpose of the study is to evaluate in novice surgeons the accuracy of the X-Guide® navigation system (X-Guide®, X-Nav Technologies®, Pennsylvania, USA) in implant placement compared to freehand implant placement.

DETAILED DESCRIPTION:
Randomized clinical trial with 2 parallel treatment groups. Eligible patients will be randomized with a 1:1 ratio to one of 2 possible parallel treatment groups:

* Group 1: Nobel Replace Conical Connection® placed freehand.
* Group 2: Nobel Replace Conical Connection® placed using the X-Guide guided surgery system (X-Nav Technologies®, Pennsylvania, USA).

PRIMARY OBJECTIVE:

- To evaluate in novice surgeons the accuracy of the X-Guide® Navigation System (X-Guide®, X-Nav Technologies®, Pennsylvania, USA) in implant placement compared to freehand implant placement.

SECONDARY OBJECTIVES:

* To evaluate overall surgical time with the X-Guide® Navigation System (X-Guide®, X-Nav Technologies®, Pennsylvania, USA) compared to freehand implant placement in inexperienced surgeons.
* To evaluate Patient Reported Outcomes Measures (PROMs) during implant treatment with navigation systems performed by novice surgeons.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who agree to voluntarily sign the informed consent before performing any action related to the study.
* Men or women at least 18 years old.
* Single edentulous spaces or edentulous sections located in maxilla or mandible with a healing period longer than 12 weeks to rehabilitate with implant-supported fixed crowns ≤3 units.
* O'Leary plaque and/or bleeding on probing index ≤25%.

Exclusion Criteria:

* Systemic diseases that may interfere with dental implant placement.
* Any contraindications for oral surgical procedures.
* History of head and neck radiotherapy.
* Patients smoking >20 cigarettes/day or tobacco equivalents.
* History of substance abuse (drugs or alcohol) or any other factor (e.g., severe psychiatric illness) that, in the opinion of the investigator, could interfere with the patient's ability to cooperate and comply with the study.
* Patients who have participated in a clinical trial within the last 30 days.
* Pregnant or lactating women.
* Patients with poor or unmotivated oral hygiene.
* Probing depth with bleeding of ≥4 mm in one of the teeth adjacent to the edentulous space or tract.
* Need to perform guided bone regeneration procedures simultaneous to implant placement.
* Cases where the use of transepithelial abutments is not recommended (reduced prosthetic space, high esthetic demand associated with thin gingival biotypes, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-09-08 (Actual); Primary Completion 2024-07-16 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
To evaluate in novice surgeons the accuracy of the X-Guide® navigation system (X-Guide®, X-Nav Technologies®, Pennsylvania, USA) in implant placement compared to freehand implant placement. | Through study completion, an average of 1 year.
  The accuracy of placement of Nobel Replace Conical Connection® implants (Nobel Biocare) will be evaluated by superimposing the two cone-beam computed tomography (CBCT) (pre- and post-surgical) and calculating the deviations from the pre-operative planning and the final implant position. The superimposition of both CBCTs will be performed using X-Guide Standalone Planning Software (Nobel Biocare).
  The following variables will be analyzed for each implant: Angular deviation, Lateral platform deviation (2D), Global platform deviation (3D), Lateral apex deviation (2D), Apex depth deviation and Global apex deviation (3D).

SECONDARY OUTCOMES:
To evaluate overall surgical time with the X-Guide® Navigation System (X-Guide®, X-Nav Technologies®, Pennsylvania, USA) compared to freehand implant placement in inexperienced surgeons. | During the surgical procedure.
  Duration of the operation from the moment of anesthesia to the last suture point. In seconds (s).
Comparison of Patient Reported Outcomes Measures (PROMs) between navigated and freehand surgery, using the Oral Health Impact Profile questionnaire, in addition to a PROMs questionnaire designed. | The OHIP-14 will be performed just before starting the surgery and at the 7-day postoperative control. The PROMs questionnaire will be performed by the patient just after finishing the implant surgery and having explained the postoperative instructions.
  A questionnaire has been designed to evaluate the PROMs of patients treated with dynamic guided surgery and compare it with the PROMs of patients treated freehand:
  * Prior to surgery the patient will complete the oral health impact profile questionnaire (OHIP-14sp).
  * Immediately after the surgery and after explaining the postoperative instructions, the patient will fill in the questionnaire designed to evaluate PROMs.
  * At 7 postoperative days, the patient will again complete the OHIP-14sp.
Comparison of postoperative pain between navigated and freehand surgery, using a questionnaire designed with a visual analog scale (VAS). | The postoperative pain will be evaluated immediately after the surgery with a VAS questionnaire and during the 7 days following surgery.
  A questionnaire has been designed to evaluate the postoperative pain of patients treated with dynamic guided surgery and compare it with patients treated freehand:
  * Immediately after the surgery the patient will complete the VAS questionnaire.
  * Another VAS questionnaire will be given to assess postoperative pain during the 7 days following surgery.
    * The VAS questionnaire consists of a 100 mm visual analog scale (VAS). In the VAS questionnaire given for the 7 postoperative days there will be a VAS for each day and the analgesics and anti-inflammatory drugs consumed by the patient will be recorded.
    * The VAS is formed by the value "No pain" to the left of the 100 mm straight line and by the value "Worst pain imaginable" to the right of the 100 mm straight line.

CONTACTS AND LOCATIONS:
Overall Officials: Eduard Valmaseda Castellón, PhD, Study Chair — University of Barcelona
Locations (1):
- University of Barcelona, L'Hospitalet de Llobregat, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No
Patients' personal data will not be published, however, the results of the scientific study will be published in a scientific dental journal.

REFERENCES:
- [Background] D'haese J, Ackhurst J, Wismeijer D, De Bruyn H, Tahmaseb A. Current state of the art of computer-guided implant surgery. Periodontol 2000. 2017 Feb;73(1):121-133. doi: 10.1111/prd.12175. PMID 28000275
- [Background] Block MS, Emery RW. Static or Dynamic Navigation for Implant Placement-Choosing the Method of Guidance. J Oral Maxillofac Surg. 2016 Feb;74(2):269-77. doi: 10.1016/j.joms.2015.09.022. Epub 2015 Sep 30. PMID 26452429
- [Background] Gaggl A, Schultes G, Karcher H. Navigational precision of drilling tools preventing damage to the mandibular canal. J Craniomaxillofac Surg. 2001 Oct;29(5):271-5. doi: 10.1054/jcms.2001.0239. PMID 11673921
- [Background] Wang F, Wang Q, Zhang J. Role of Dynamic Navigation Systems in Enhancing the Accuracy of Implant Placement: A Systematic Review and Meta-Analysis of Clinical Studies. J Oral Maxillofac Surg. 2021 Oct;79(10):2061-2070. doi: 10.1016/j.joms.2021.06.005. Epub 2021 Jun 10. PMID 34245701
- [Background] Pellegrino G, Ferri A, Del Fabbro M, Prati C, Gandolfi MG, Marchetti C. Dynamic Navigation in Implant Dentistry: A Systematic Review and Meta-analysis. Int J Oral Maxillofac Implants. 2021 Sep-Oct;36(5):e121-e140. doi: 10.11607/jomi.8770. PMID 34698720
- [Background] Jorba-Garcia A, Gonzalez-Barnadas A, Camps-Font O, Figueiredo R, Valmaseda-Castellon E. Accuracy assessment of dynamic computer-aided implant placement: a systematic review and meta-analysis. Clin Oral Investig. 2021 May;25(5):2479-2494. doi: 10.1007/s00784-021-03833-8. Epub 2021 Feb 26. PMID 33635397
- [Background] Emery RW, Merritt SA, Lank K, Gibbs JD. Accuracy of Dynamic Navigation for Dental Implant Placement-Model-Based Evaluation. J Oral Implantol. 2016 Oct;42(5):399-405. doi: 10.1563/aaid-joi-D-16-00025. Epub 2016 Jun 6. PMID 27267658
- [Background] Jorba-Garcia A, Figueiredo R, Gonzalez-Barnadas A, Camps-Font O, Valmaseda-Castellon E. Accuracy and the role of experience in dynamic computer guided dental implant surgery: An in-vitro study. Med Oral Patol Oral Cir Bucal. 2019 Jan 1;24(1):e76-e83. doi: 10.4317/medoral.22785. PMID 30573712
- [Result] Vercruyssen M, Fortin T, Widmann G, Jacobs R, Quirynen M. Different techniques of static/dynamic guided implant surgery: modalities and indications. Periodontol 2000. 2014 Oct;66(1):214-27. doi: 10.1111/prd.12056. PMID 25123770
- [Result] Miller RJ, Bier J. Surgical navigation in oral implantology. Implant Dent. 2006 Mar;15(1):41-7. doi: 10.1097/01.id.0000202637.61180.2b. PMID 16569960

DOCUMENTS (1):
  • Informed Consent Form (2023-08-30): https://cdn.clinicaltrials.gov/large-docs/50/NCT06028750/ICF_000.pdf